CLINICAL TRIAL: NCT05056415
Title: Effect and Cost-effectiveness of the 'Everyday Life Rehabilitation' Intervention: a Pragmatic RCT of Integrated, Recovery-focused Rehabilitation Within Sheltered and Supported Housing Facilities for People With Psychiatric Disabilities
Brief Title: Effect and Cost-effectiveness of the Everyday Life Rehabilitation Intervention
Acronym: ELR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Maria Lindstrom, Principal Investigator, Assistant professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 330210302 - FORTE 2021-2024, M
Record Dates: First submitted 2021-09-04; First posted 2021-09-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psychiatric or Mood Diseases or Conditions; Neuropsychiatric Syndrome; Psychosis; Autism; Severe Mental Disorder
Keywords: RCT; effect; cost-effectiveness; equity; severe psychiatric disability; personcentered; personal recovery; Everyday Life Rehabilitation; Occupational Therapy
MeSH Terms: conditions — Psychotic Disorders; Autistic Disorder; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): In the involved municipalities, TAU mainly consists of short-term efforts, such as Occupational Therapist (OT) prescribing technical aids, often initiated by the housing staff (HS). Daily support provided by HS varies, depending on the approach and commitment of individual staff and the norms that prevail in different housing units, as well as variations between municipalities. Co-planning on long-term rehabilitation efforts does not exist or is weak, and collaboration between OT and HS is, as described by staff from both parties, difficult to achieve.
  After a control-period of 6 month, house facilities within the TAU-group will also be offered ELR.
  Interventions: Other: Treatment as usual (TAU)
- Everyday Life Rehabilitation (ELR) plus TAU (Experimental): ELR is a model for long-term, outreach, and personalized rehabilitation for persons with SPD living in sheltered or supported housing facilities, in close collaboration between resident, OT, and HS.
  ELR includes personcentred, motivational-, recovery- and activity-based methods, built on certain process steps. The focus is to promote personal recovery, while targeting meaningful daily activities, through person-driven goals, negotiated expectations, exploration and activity-training in real-life situations, and a maintenance phase. ELR includes a web-based educational package, and devices for reflective collaborative learning.
  ELR consists of a weekly session with an OT, followed by regular collaboration with HS, who support the resident on a daily basis, in line with guidance given by the OT and input shared from the HS. The intervention period will last for 6 months.
  Prior to the intervention, OT, HS, and HM will partake in web-based training, with associated manuals, and tools.
  Interventions: Other: Everyday Life Rehabilitation (ELR)

INTERVENTIONS:
Other: Everyday Life Rehabilitation (ELR) — Everyday Life Rehabilitation (ELR) is an intervention model for integrated occupational therapy in close collaboration with housing staff in sheltered and supported housing facilities (Lindström, 2007; 2011), aiming at personal recovery and engagement in meaningful everyday activities for persons with SPD. The mediators are: personcentred, motivational, recovery- and activity-based methods, negotiation of user goal priority and expected outcome; methods for training in real-life situations; devices for collaboration; support from staff on an everyday basis; and an educational package including web-sections, manuals, and collegiate tutorial.
  The language and actions of professionals promote hope, self-discovery and shared-decision making, shaped in partnership with residents. The resident is also encouraged to access different resources outside of health and social care such as family, peer and social support, out-of-housing strategies, and sources in the open society.
  Arms: Everyday Life Rehabilitation (ELR) plus TAU
Other: Treatment as usual (TAU) — No standardized instructions about the efforts is given to staff at the accommodations. Usually, only short terms efforts are offered to residents, such as prescribing technical aids.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The person-centered, motivational, recovery-, and activity-based intervention model 'Everyday Life Rehabilitation´ (ELR), integrated in sheltered and supported housing facilities for people with severe psychiatric disabilities, has shown significant outcomes in feasibility studies, and thus a RCT is required, for the purpose of establishing the effectiveness and cost-effectiveness of ELR.

All municipalities in northern and middle Sweden will be invited. Residents who meet the inclusion criteria, will be invited to participate. Housing-units, with associated residents giving consent, will be randomized to either receive intervention with ELR plus treatment as usual (TAU), or TAU alone for control group. Hence, the present study is a cluster RCT. The control group will, after control-period, be offered ELR. Professionals involved in the ELR intervention group; that is occupational therapists, housing staff and housing managers, will receive an educational package. It is hypothesized that the intervention-group will improve in personal and social recovery as well as quality of life.

The primary outcome is recovering quality of life assessed by ReQoL, and secondary outcomes are self-perceived recovery, everyday functioning, and goal-attainment at 6 months, assessed using RAS-DS, and GAS, respectively. ReQoL will be transformed into QALY´s for calculation of cost-effectiveness.

The study has an adaptive design, including an internal pilot year one and two, in order to determine required sample sizes before continuing with the full scale RCT.

DETAILED DESCRIPTION:
The investigators intend to study the extent to which the intervention under study; the Everyday Life Rehabilitation (ELR), is an effective, and cost-effective model for co-planned rehabilitative services in sheltered and supported housing facilities, aiming at supporting residents´ personalized recovery pathway. The project is of high relevance with its permeating perspectives of severe psychiatric disability (SPD), equity, and quality improvement, in the intersection of health and social care in accommodations.

The ELR project is both user- and practice-oriented. The main focus is to study whether the ELR-model is effective, cost-effective, and relevant for users, based on pre-/post-intervention variables from a resident perspective, such as self-perceived recovery, quality of life, everyday functioning, and goal fulfilment of residents. The project is also practice-oriented with a web-based training, methods and tools for staff. The project is pragmatic in the sense of implementing and studying the ELR model in as natural context as possible. Throughout the investigators will collaborate with user- and relative associations, municipalities, and R&D units, in order to develop an intervention that is relevant and useful.

It has been shown that people with SPD and impaired autonomy have significantly poorer health than the general population, while at the same time they do not have access to equal health care, despite that they belong to the highest priority group according to the Swedish Parliament's principles for prioritization of healthcare. The high priority is based on the fact that the target group has low autonomy and does not speak out loudly for themselves, or can argue for their right to health care, further that they do not actively seek and demand health care, along with the magnitude of suffering, and the impact on life quality. There is a gap in knowledge, regulations, and lack of interventions suiting this context. Both rehabilitative healthcare interventions in practice, and RCT´s, are sparse regarding interventions for this target group living in sheltered or supported housing facilities. Thus, it is important to develop and test new potentially useful and effective interventions.

Therefore, a manualized but individually flexible model for integrated healthcare-rehabilitation in collaboration with housing staff in supported or sheltered housing facilities; the Everyday Life Rehabilitation (ELR), has been developed by the project manager (Lindström, 2007), and tested in feasibility studies (Lindström et al, 2011; 2011b; 2012; 2013; 2017), aiming at personal recovery and meaningful everyday activities for persons with SPD. The ELR development is thus based on five years of previous research with feasibility studies, and has shown significant impact on residents' everyday functioning and health, as well as the practices of professionals. Based on these feasibility studies, the original ELR has been slightly revised, adding a monthly follow-up by housing managers, and clarified tools for co-planning, in order to promote early involvement in enhancing strategies. The Medical Research Council (MRC) guidelines for complex interventions have been thoroughly applied in the development process, and next, evidence is needed for implementation, requiring randomized controlled trial (RCT)-studies. Therefore, the investigators want to expand the design, and go further with a cluster RCT built on a slightly revised manual of the ELR intervention, adding clarified focus on management, the tools for collaboration, and a cost-effectiveness perspective.

Overall aim and research questions:

The overall aim of the project is to investigate the effectiveness, and cost-effectiveness of a co-planning, person-centered, motivational, recovery-, and activity-based intervention package for people with SPD living in sheltered or supported housing facilities.

The specific research questions (RQs) are as follows 1-2:

RQ 1. What is the effectiveness of ELR intervention on recovery, quality of life, everyday functioning, and goal attainment, compared to Treatment as usual (TAU)? RQ 2. What is the estimated cost-effectiveness based on participant outcomes following ELR plus TAU, and TAU alone, according to baseline differences of recovering quality of life (ReQoL) transformed into QALY´s? For RQ 1 and 2, data will be collected pre- and post intervention. Allocation will be concealed for the independent blinded testers, and partly concealed for the people with SPD giving consent to participate in the study, being informed that a waiting list of up to six months may become relevant. The treating occupational therapists, housing staff, and housing managers, will due to practical reasons not be masked to the intervention. Data will also be blinded to researchers until analysis have been conducted. A person at Umeå university, who is not involved in neither the interventions nor analysis, will administrate, collect and store coded data in a safety-box.

An initial power-analysis was conducted, dimensioning the study to detect a difference of 5 points on the ReQoL-scale with 80% power. Assuming a standard deviation of 10 (Keetharuth et al, 2018), an average cluster size of 2 participants per hosting facility and an intraclass correlation of 0.1, a total of 35 housing facilities in each group is required to reach a power of 80% when using a significance level of 5%.

Oral explanation of the study and a leaflet describing the methods will be given prior to the participant consent. Considering the target population of the intervention is a vulnerable group, there are particular ethical reasons to minimize the number of exposed participants, and thus an internal pilot from year one and two will form the basis for the determination of the sample size for the full scale RCT. This is in line with the recommendation of MRC guidelines for complex intervention.

Statistical analyses:

Regarding analysis for RQ 1, mixed effects models will be used to analyse the primary outcome, including a random intercept for the clustering factor housing facility. The post-intervention measurements will be used as outcome variables, while adjusting for corresponding baseline measurements. The adjustment for baseline variables will performed on both individual level and on aggregated cluster level using the average of the baseline measurement within the housing facility (Hooper et al, 2018). Details about the model, and the adjustment for baseline covariates will be prespecified in thein the statistical analysis plan.

The primary analysis will use an intention-to-treat (ITT) approach and include all allocated participants with valid data, whether they did or did not receive the complete intervention. Multiple imputation will be used for variables where missing-at-random can be assumed. A complementary per protocol analysis will also be made.

For the intervention group only, goal attainment scaling (GAS) will be calculated according to the specific statistical formula of GAS. The secondary outcomes (RAS-DS and GAS) will be analysed using mixed effects models or semi-parametric ordinal cumulative link models, including housing facility as a random effect. This is pre-specified in detail in the statistical analysis plan.

Subgroup analysis will also be conducted, stratifying on gender in all outcomes.

Specifically, for RQ2 on cost-effectiveness, the following analyses will be conducted: For univariate testing of significance of cost and ReQoL, Student´s test will initially be used. For cost-effectiveness analysis, the costs and effects of the ELR and the TAU alternative, will be calculated and presented in a ratio of incremental cost to incremental effect. Effects are health outcomes, such as quality-adjusted-life-years (QALY). For this matter, ReQoL will be transformed into QALY, accounting for baseline differences.

The Swedish Board for Health and Welfare has developed a model for priorities in health care, which consists of the following criteria: severity of the condition, effectiveness in treatment, cost-effectiveness in treatment, and evidence base. The model assumes a specific condition linked to a specific treatment.

In this study the conditions are X and Y, and the treatments are X and Y. This study is designed to provide this model with proper data. A high degree of severity in these conditions have repeatedly been reported.

Thus, the trial is designed to measure effectiveness, and cost-effectiveness. The latter is defined as the cost per QALY gained. The resources needed for the interventions will be measured in physical units (mainly time) and transformed to monetary values.

When all sub-studies have been finalized, the investigators plan to suggest a priority rank for the interventions under study. The Board for Health and Welfare use a scale in 10 steps; 1 is the highest possible rank and 10 is the lowest. This ranking is based on the four criteria described above.

Protocol amendments:

After the first year, the internal pilot will be analyzed. A non-comparative interim analysis will be performed to assess variability in outcome variables. This will form the basis of an updated sample size calculation.

The internal pilot will also be used as a basis for possible minor adjustments of the study protocol. In addition, feasibility of the full scale study will be evaluated. Should it be concluded that ethical problems arise due to unexpected problems in the study process and it is unlikely that further knowledge will be gained from continuing the full study with recruitment of more housing facilities and participants, the study will be interrupted. Results and gained insights about feasibility from the interval pilot alone will be published.

Results and conclusions from the internal pilot will be presented at the trial's site at clinicaltrials.gov. Any adjustments of the protocol and the statistical analysis plan following from the evaluation of the internal pilot will be published as amendments.

3-year update: the recruitment was somewhat slower than expected, and sample size recalculation based on data from the internal pilot showed that the original target sample size would render in an expected statistical power of 53% for detecting a group difference of 5 points in ReQoL. Therefore, the investigators decided to redimension the study to detect a group difference of 10 points, which has been pointed out as a minimum clinically important difference for ReQoL by the instrument developers. Given that the expected number of recruited housing units will be 45, revised calculations based on Monte Carlo simulations showed that this should be sufficient to reach 80% for detecting a group difference of 10 points. Descriptions of the sample size calculations are available in the statistical analysis plan.

ELIGIBILITY:
Inclusion criteria:

* adults with severe psychiatric disability (SPD)
* living in sheltered or supported housing facility for people with SPD in municipalities within the geografic area and with access to occupational therapy

Exclusion criteria:

* comorbidity of dementia or severe developmental disability
* not being able to communicate in Swedish
* currently being in acute psychosis, or acute suicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline 'Recovering quality of life score' at 6 months | Measurements will be conducted pre-, and post intervention-/control-period of six months
  Recovering quality of life will be measured for RQ 1 and RQ 2 using the Recovering quality of life (ReQoL) (Keetharuth et al, 2018).
  ReQoL applies to the whole spectrum of mental health conditions, from common mental health disorders through to very severe ones.
  ReQoL are comprised of positive and negative worded items. Items cover areas of quality of life, shown to be important for service users: Activity (meaningful); Belonging and relationships; Choice, control and autonomy; Hope; Self-perception; Well-being; and Physical health.
  An increase of points on the ReQoL score denotes improvement. In ReQoL-20, the minimum score is 0 and the maximum is 80, where 0 indicates poorest quality of life and 80 indicates highest quality of life. Preference weights are available for the ReQoL to generate quality adjusted life years (QALYs).

SECONDARY OUTCOMES:
Change from baseline 'Total Recovery score' at 6 months | Measurements will be conducted pre-, and post intervention-/control-period of six months
  Secondary outcome for RQ1 is self-perceived personal recovery and daily functioning, assessed using the Recovery Assessment Scale - Domains & Stages (RAS-DS) (Hancock et al, 2016). A total recovery score is gained from adding the scores for all items. The maximum score is 152.

OTHER OUTCOMES:
Goal Attainment at 6 months | Goal attainment will be measured after an intervention-period of six months.
  Goal-attainment will be measured within the intervention group only, using the Goal Attainment Scaling (GAS) (Kiresuk et al, 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lindström, PhD, Principal Investigator — Umeå university, Dept of Community Medicine and Rehabilitation
Locations (1):
- Umeå university, Umeå, Sweden

REFERENCES:
- [Derived] Sjoberg A, Liv P, Lindstrom M. Effect of Everyday Life Rehabilitation on recovering quality of life in individuals with serious mental illness in supported accommodation: a pragmatic cluster randomised controlled trial. BMJ Ment Health. 2025 Aug 7;28(1):e301757. doi: 10.1136/bmjment-2025-301757. PMID 40780841
- [Derived] Lindstrom M. Development of the Everyday Life Rehabilitation model for persons with long-term and complex mental health needs: Preliminary process findings on usefulness and implementation aspects in sheltered and supported housing facilities. Front Psychiatry. 2022 Aug 16;13:954068. doi: 10.3389/fpsyt.2022.954068. eCollection 2022. PMID 36051549
- [Derived] Lindstrom M, Lindholm L, Liv P. Study protocol for a pragmatic cluster RCT on the effect and cost-effectiveness of Everyday Life Rehabilitation versus treatment as usual for persons with severe psychiatric disability living in sheltered or supported housing facilities. Trials. 2022 Aug 15;23(1):657. doi: 10.1186/s13063-022-06622-0. PMID 35971130

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05056415/SAP_001.pdf